CLINICAL TRIAL: NCT07383103
Title: Initiation of Hydrocortisone and Fludrocortisone in Adult Patients With Septic Shock：A Prospective Randomized Controlled Clinical Trial
Brief Title: Hydrocortisone and Fludrocortisone for the Treatment of Septic Shock
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Qing-quan Lv, Principal Investigator, Northern Jiangsu People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025ky387
Record Dates: First submitted 2026-01-25; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Septic Shock
Keywords: septic shock; hydrocortisone; fludrocortisone; mortality
MeSH Terms: conditions — Shock, Septic | interventions — Hydrocortisone; Fludrocortisone; fludrocortisone acetate; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrocortisone plus Fludrocortisone (Experimental): Hydrocortisone: 200 mg per day administered by continuous intravenous infusion for up to 7 days or until ICU discharge, whichever occurs first.
  Fludrocortisone: 50 μg administered orally or via nasogastric tube once daily for up to 7 days or until ICU discharge, whichever occurs first.
  Interventions: Drug: Hydrocortisone plus Fludrocortisone
- Standard care (Active Comparator): Patients will receive standard care for septic shock according to current international guidelines, including fluid resuscitation, vasopressor therapy, antimicrobial treatment, and other supportive measures, including the use of hydrocortisone at the discretion of the treating physician, but without fludrocortisone.
  Interventions: Other: Standard care

INTERVENTIONS:
Drug: Hydrocortisone plus Fludrocortisone — Hydrocortisone will be administered at a dose of 200 mg per day by continuous intravenous infusion.
  Fludrocortisone will be administered at a dose of 50 μg once daily orally or via nasogastric tube.
  Both drugs will be given for up to 7 days or until ICU discharge, whichever occurs first.
  Other Names: Hydrocortisone Injection; Fludrocortisone Acetate Tablets
  Arms: Hydrocortisone plus Fludrocortisone
Other: Standard care — Patients will receive standard care for septic shock according to current international and institutional guidelines, including fluid resuscitation, vasopressor therapy, antimicrobial treatment, and other supportive measures. Fludrocortisone will not be administered.Hydrocortisone may be administered at the discretion of the treating physician.
  Arms: Standard care

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the combination therapy of hydrocortisone and fludrocortisone among adult patients with septic shock.

DETAILED DESCRIPTION:
Sepsis is a life-threatening organ dysfunction caused by a dysregulated host response to infection, and septic shock represents its most severe form, characterized by profound circulatory and metabolic abnormalities with high mortality.

Current international guidelines recommend intravenous hydrocortisone as adjunctive therapy in patients with septic shock who remain hypotensive despite adequate fluid resuscitation and vasopressor treatment. However, critically ill patients may exhibit relative deficiencies of both glucocorticoid and mineralocorticoid activity, and hydrocortisone alone may not fully meet the physiological demands under severe stress. In recent years, combination therapy with hydrocortisone and fludrocortisone has been investigated, but published trials have reported inconsistent results regarding mortality, shock reversal, and adverse events.

Therefore, this randomized controlled trial aims to evaluate the efficacy and safety of hydrocortisone combined with fludrocortisone, compared with standard therapy, in patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

(1)18≤Age≤90; (2)Diagnosis of septic shock within 12 h.

Exclusion Criteria:

Patients meeting any of the following conditions will be excluded:

1. Systemic corticosteroid therapy within the last 3 months before septic shock;
2. High-dose steroid therapy;
3. Immunosuppression;
4. Pregnant;
5. Known allergy to hydrocortisone or fludrocortisone;
6. Presence of gastrointestinal bleeding, perforation, or other conditions requiring fasting;
7. Anticipated death from a preexisting disease within 90 days after randomization (as determined by the enrolling physician);
8. Refusal of the attending staff or patient family;
9. Current participation in another clinical trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
90-day mortality | 90 days after randomization
  All-cause mortality at day 90 after randomization

SECONDARY OUTCOMES:
28-day mortality | 28 days after randomization
  All-cause mortality at day 28 after randomization
ICU mortality | From randomization to ICU discharge (up to 90 days)
  All-cause mortality at ICU discharge
Hospital mortality | From randomization to hospital discharge (up to 90 days)
  All-cause mortality at hospital discharge

OTHER OUTCOMES:
Shock reversal time | From randomization up to 28 days
  Reversal of shock is defined as the maintenance of a systolic blood pressure of at least 90 mmHg without vasopressor support for at least 24 h. Time to shock reversal is defined as the time from randomization to shock reversal.
ICU length of stay | From randomization to ICU discharge (up to 90 days)
  Time in days until ICU discharge
Hospital length of stay | From randomization to hospital discharge (up to 90 days)
  Time in days until hospital discharge
Change in Sequential Organ Failure Assessment (SOFA) score at 72 hours | 72 hours after randomization
  The Sequential Organ Failure Assessment (SOFA) score ranges from 0 to 24, with higher scores indicating more severe organ dysfunction and worse clinical outcomes. The change in SOFA score (ΔSOFA) is calculated as the SOFA score at enrollment minus the SOFA score at 72 hours after randomization. If a patient is discharged from the ICU within 72 hours, the SOFA score at ICU discharge will be used for analysis.
72h lactate | 72 hours after randomization
  lactate level at 72h after randomization
72h P/F | 72 hours after randomization
  P/F at 72h after randomization
ICU-free days up to day 28 | 28 days after randomization
  Total number of days alive and free of ICU stay during the 28 days after randomization.
Vasopressor-free days up to day 28 | 28 days after randomization
  Total number of days alive and free of vasopressor during the 28 days after randomization.
Ventilator support-free days up to day 28 | 28 days after randomization
  Total number of days alive and free of ventilator support during the 28 days after randomization.
CRRT-free days up to day 28 | 28 days after randomization
  Total number of days alive and free of CRRT during the 28 days after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Qingquan Lyu, Master, Principal Investigator — Northern Jiangsu People's Hospital
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No